CLINICAL TRIAL: NCT04280172
Title: Educational Intervention to Support Development of Mentors' Cultural Competence and Competence in Mentoring Culturally and Linguistically Diverse Nursing Students
Brief Title: Effectiveness of Cultural Competence Education for Nurse Mentors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: The Finnish Association of Nursing Research (Unknown); Finnish Nurses Association (Unknown)
Responsible Party: Principal Investigator, Ashlee Oikarainen, Researcher, University of Oulu
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CulturalCompetence
Record Dates: First submitted 2020-02-13; First posted 2020-02-21 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Cultural Competency; Mentoring

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cultural Competence Education (Experimental): Participants in the intervention group will attend cultural competence education
  Interventions: Other: Cultural Competence Education
- Standard Mentoring Education (Active Comparator): Participants in the control group will complete standard mentoring education that does not include a cultural competence component
  Interventions: Other: Standard Mentoring Education

INTERVENTIONS:
Other: Cultural Competence Education — Cultural competence education for participants in the intervention group comprises of completion of an online learning module and participation in an eight-hour training day. The educational content includes various topics related to cultural and linguistic diversity and cultural competence in mentoring.
  Arms: Cultural Competence Education
Other: Standard Mentoring Education — Participants in the control group will not receive the educational intervention but will participate in standard mentoring education. This education is offered in an online learning environment and participants can complete the education at their own pace. The educational content focuses on general issues related to mentoring and does not contain topics specific to cultural competence in mentoring.
  Arms: Standard Mentoring Education

SUMMARY:
Clinical placements are an integral part of nursing education and have significant impact on nursing students' professional development. According to standards set by the European Union, the duration of clinical placements should account for at least one half of the minimum duration of nursing programs. Also, students must complete training under the supervision of qualified nursing staff (Directive 2013/55/EU of the European Parliament and of the Council).

Nursing staff are responsible for the mentoring of students during completion of their clinical placements. The role of the mentor can be challenging and several studies prove that providing continuing education to mentors can be effective in developing mentors' competence in mentoring. There is an urgent need to add issues related to the development of mentors' cultural competence into mentoring education. This is due to the rapid increase of cultural and linguistic diversity within the nursing workforce and the increase in the numbers of students from international backgrounds.

This study is designed to assess the effectiveness of an educational intervention to develop mentors' cultural competence and their competence in mentoring nursing students from diverse cultural and linguistic backgrounds.

DETAILED DESCRIPTION:
METHODOLOGY

Study setting:

The study will be conducted in two hospitals, which are located in two different major cities in Finland.

Study design:

This is a nonrandomized, pre-post quasi-experimental study. Participants in this study will participate in cultural competence education. Participants will self-assess their level of competence in mentoring in general along with their cultural competence in mentoring. There will be three assessment time points: at baseline (before education, T0), immediately after the education (T1), and 6 months after the education (T2). The control group will receive standard mentoring education that does not contain topics specific to cultural competence or the mentoring of students from diverse backgrounds. The same self-assessment instrument and assessment time points will be used for both the intervention and control groups.

Study size:

A total of 60 mentors will be allocated to the intervention group and 60 mentors to the control group.

Study duration:

The educational intervention (cultural competence education) will be conducted for a duration of 9 months (T0, T1, T2). The education will be offered twice (fall 2020, spring 2021), thus the total duration of the study (from date study open for recruitment to final data collection) will be a total of 16 months.

Sampling of participants

Recruitment:

Participants in the intervention group who attend cultural competence education and participants who belong to the control group will be recruited into this study via internal recruitment methods implemented by clinical coordinators employed at the participating hospitals.

Intervention:

Cultural competence education for participants in the intervention group comprises of completion of an online learning module and participation in an eight-hour training day. The educational content includes various topics related to cultural and linguistic diversity and cultural competence in mentoring.

Control:

Participants in the control group will not receive the educational intervention but will participate in standard mentoring education offered at the participating university hospital. This education is offered in an online learning environment and participants can complete the education at their own pace. The educational content focuses on general issues related to mentoring and does not contain topics specific to cultural competence in mentoring.

Sample size

A power analysis has been calculated for an effect size according to Cohen's d, two tail-test, significance at p<0.05, power of 80% (1- Beta err prob). The estimated sample size was 60 participants per group after accounting for significance level of 0.05%, power of 80% and 50% attrition.

INSTRUMENTS AND DATA COLLECTION

Intervention: Cultural competence education

Questionnaire: Mentors' competence in mentoring will be measured using the psychometrically validated self-assessment Mentors' Competence Instrument (MCI). A newly developed Mentors' Cultural Competence Instrument (MCCI) will be used to measure mentors' cultural competence. This instrument has been administered and pilot tested by 12 mentors prior to implementation of the intervention.

Finnish language versions of the questionnaire will be administered containing the following sections:

1. Sociodemographic data:

   * Sex
   * Age
   * Educational background
   * Place of work
   * Current position
   * Work experience
   * Name of work organization
   * Current work unit
   * Time when last mentored a student
   * Time used for reflective discussion with student
   * Previous participation in mentoring education
   * Experience mentoring international students
   * How often international students are mentored
2. Competence in mentoring using Mentors' Competence Instrument which contains 43 items divided into 7 sections

   * Mentoring practices between the student and mentor
   * Mentor's characteristics
   * Mentor's motivation
   * Goal-oriented mentoring
   * Reflection during mentoring
   * Student-centered evaluation
   * Constructive feedback
3. Mentors' cultural competence using Mentors' Cultural Competence Instrument which contains 21 items covering the following topics

   * Cultural sensitivity and awareness
   * Cultural knowledge
   * Intercultural communication and interaction
   * Cultural skills and safety

DATA COLLECTION

Intervention group

1. Baseline questionnaire (T0): Paper-based questionnaires will be administered to participants in the intervention group on the day of study recruitment before being given details on how to complete the cultural competence education.
2. Post course questionnaire (T1): Paper-based questionnaires will be administered to participants in the intervention group immediately following completion of the cultural competence education.

   a. Participants will be asked to provide their evaluation of the education in addition to the questionnaire described above. The evaluation contains the following questions:
   * How satisfied were you with the mentoring education?
   * Did the mentoring education have an impact on your ability to mentor students?
   * Did the mentoring education have an impact on your willingness to mentor students?
   * Open comment section for comments or concerns regarding the mentoring education
3. 6-month follow up questionnaire (T2): Paper-based questionnaires including will be sent to participants via post to participants' home addresses.

Control group

1. Baseline questionnaire (T0): Web-based questionnaires will be administered to participants in the control group on the first day of standard online mentoring education.
2. Post course questionnaire (T1): Web-based questionnaires will be administered to participants in the control group on the last day of standard online mentoring education.
3. 6-month follow up questionnaire (T2): Web-based questionnaires will be sent to participants via email six months following completion of the standard online mentoring education.

ETHICAL CONSIDERATIONS This study complies with the standards and guidelines of the responsible conduct of research. The necessary research permissions from the participating hospitals have been obtained prior to data collection and implementation of the intervention. In this study, formal approval from an ethics committee is not required. Participation is voluntary and participants will be informed of the purpose of the study and their right to withdraw from the study. Participants' confidentiality and anonymity will be protected and research data will be secured according to current standards.

Data analysis Data will be analyzed using IBM Social Package for Social Science (SPSS, version 26). Data will be analyzed using descriptive statistics, a Wilcoxon Signed-Rank Test and a two-way ANOVA test. In this study, two-tailed testing will be used and the significance level will be set at a p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* be currently employed in any professional nursing role on any unit; have the skills to read and understand the Finnish language; and consent to participate in the study

Exclusion Criteria:

- be on long-term leave of absence or maternity leave; lack of skills to read and understand the Finnish language, decline to consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in mentors' cultural competence | Pre intervention, immediately after intervention and 6 months after intervention
  Mentors' cultural competence will be measured using the newly developed Mentors' Cultural Competence Instrument. The instrument contains 21 items using a four-level Likert scale. A higher score on the likert scale indicates a higher level of competence.
Changes in competence in mentoring | Pre intervention, immediately after intervention and 6 months after intervention
  Mentors' competence in mentoring will be measured using the psychometrically validated self-assessment Mentors' Competence Instrument (MCI), which contains 43 items divided into 7 sections using a four-level Likert scale. A higher score on the Likert scale indicates a higher level of competence.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Mikkonen, PhD, Study Chair — University of Oulu; Ashlee I Oikarainen, MHSc, Principal Investigator — University of Oulu
Locations (2):
- Finland (2):
  - Healthcare organization in eastern Finland, Kuopio
  - Healthcare organizations in Nordic Finland, Oulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oikarainen A, Mikkonen K, Tuomikoski AM, Elo S, Pitkanen S, Ruotsalainen H, Kaariainen M. Mentors' competence in mentoring culturally and linguistically diverse nursing students during clinical placement. J Adv Nurs. 2018 Jan;74(1):148-159. doi: 10.1111/jan.13388. Epub 2017 Aug 1. PMID 28702955
- [Background] Oikarainen A, Mikkonen K, Kenny A, Tomietto M, Tuomikoski AM, Merilainen M, Miettunen J, Kaariainen M. Educational interventions designed to develop nurses' cultural competence: A systematic review. Int J Nurs Stud. 2019 Oct;98:75-86. doi: 10.1016/j.ijnurstu.2019.06.005. Epub 2019 Jun 21. PMID 31319338
- [Derived] Oikarainen A, Kaarlela V, Heiskanen M, Taam-Ukkonen M, Lehtimaja I, Karsamanoja T, Tuomikoski AM, Kaariainen M, Tomietto M, Mikkonen K. Educational intervention to support development of mentors' competence in mentoring culturally and linguistically diverse nursing students: A quasi-experimental study. Nurse Educ Today. 2022 Sep;116:105424. doi: 10.1016/j.nedt.2022.105424. Epub 2022 May 29. PMID 35714426